CLINICAL TRIAL: NCT01807260
Title: STEPWISE SHOCK WAVE LITHOTRIPSY IN PEDIATRIC UROLITHIASIS: A COMPARATIVE STUDY.
Brief Title: Stepwise Shock Wave Lithotripsy in Pediatric Urolithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Assistant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: stepwise0946
Record Dates: First submitted 2013-02-28; First posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Pediatric Urinary Lithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional Shock wave lithotripsy group (Active Comparator): All procedures were performed under continu¬ous intravenous sedo-analgesia (using a combi-nation of ketamine 1 mg/kg and propofol 0,5-1 mg/kg) with fluoroscopic or ultrasonograpic imaging in a supine position. Shock wave number was limited to a maximum of 3000 waves/session. In the conventional group the voltage was only 13 kV. The stone burden was defined as the stone area that was calculated by multiply¬ing the largest length and width of the individual stones measured from the abdominal plain X-ray.
  Interventions: Procedure: Shock wave lithotripsy
- stepwise Shock wave lithotripsy group (Active Comparator): All procedures were performed under continu¬ous intravenous sedo-analgesia (using a combi-nation of ketamine 1 mg/kg and propofol 0,5-1 mg/kg) with fluoroscopic or ultrasonograpic imaging in a supine position. Shock wave number was limited to a maximum of 3000 waves/session. In the stepwise group, the voltage was started at 10 kV and increased stepwise (every 250 shock waves) to 13 kV. The stone burden was defined as the stone area that was calculated by multiply¬ing the largest length and width of the individual stones measured from the abdominal plain X-ray.
  Interventions: Procedure: Shock wave lithotripsy

INTERVENTIONS:
Procedure: Shock wave lithotripsy — All procedures were performed under continuous intravenous sedo-analgesia (using a combination of ketamine 1 mg/kg and propofol 0,5-1 mg/kg) with fluoroscopic or ultrasonograpic imaging in a supine position. Shock wave lithotrpisy was poerformed with a Dornier Compact Delta lithotripter (Dornier Medtech, Germany). Shock wave number was limited to a maximum of 3000 waves/session. In the conventional group the voltage was only 13 kV. The stone burden was defined as the stone area that was calculated by multiplying the largest length and width of the individual stones measured from the abdominal plain X-ray.

SUMMARY:
To evaluate and compare the results of conventional and stepwise shock wave lithotripsy treatment modalities in pediatric urinary lithiasis.

DETAILED DESCRIPTION:
Between March 2008 and February 2012, 81 patients were randomized and included in this study. Shock wave lithotripsy was performed by using a Dornier Compact Delta instrument. Localizations of radiopaque and non-opaque stones were estimated by using flouroscopy and ultrasonography, respectively. Treatment energy was set on 13 kV in the conventional group. In the stepwise group, treatment energy was initially set on 10 kV and gradually increased up to 13 kV per 250 shocks. The maximum numbers of shocks in both groups were limited to 3000. Patients were followed up with 15 days interval. In each visit, patients were respectively questioned for pain, hematuria and history of stone passage. In case of treatment failure, shock wave lithotripsy was repeated.

ELIGIBILITY:
Inclusion Criteria:

The patients with pediatric urinary lithiasis.

Exclusion Criteria:

Resistant urinary tract infections Coagulopathies Anatomically obstructed urinary system

Ages: 12 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2008-03; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Stone burden on plain X-ray. | Three months.
  The stone burden was defined as the stone area that was calculated by multiplying the largest length(cm)and width (cm)of the individual stones measured from the abdominal plain X-ray. To detect fragmentation of the stone and necessity of re-treatment a plain film were used during control. Stone clearance was assessed at three months. Stone-free state was defined as the absence of stone fragments on a good quality plain X-ray. Clinical success was considered if the residual fragments were 2-3 mm or less in asymptomatic patients.

OTHER OUTCOMES:
Degree and presence of hydronephrosis. | Three months
  To detect obstruction in the system, ultrasonography was used during control.
Stone burden on spiral computed tomography | Three months
  In case of non-opaque Stones, stone borden was evalusted with spinal computed tomography. Clinical success was considered if the residual fragments were 2-3 mm or less in asymptomatic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Demirci, Prof., Study Chair — Department of Urology, Erciyes University Medical faculty,
Locations (1):
- Department of Urology, Erciyes University Medical Faculty,, Kayseri, Talas, Turkey (Türkiye)

REFERENCES:
- [Result] Demirci D, Altiok E, Gulmez I, Ekmekcioglu O, Poyrazoglu HM. Stepwise shock wave lithotripsy: results of initial study for the treatment of urinary stones in childhood. Int Urol Nephrol. 2006;38(2):189-92. doi: 10.1007/s11255-005-4971-x. PMID 16868680